CLINICAL TRIAL: NCT04054713
Title: Acetic Acid vs Seattle Protocol for Neoplastic Lesions in Barrett Esophagus
Brief Title: Acetic Acid for the Detection of Esophageal Neoplasms
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients enrolled
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: R-2019-3601-143
Record Dates: First submitted 2019-07-25; First posted 2019-08-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Barretts Esophagus With Low Grade Dysplasia; Dysplasia; Intestinal Metaplasia
Keywords: Barrett Esophagus; Dysplasia; acetic acid; Seattle protocol; Chromoendoscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Intervention Model Description: A clinical trial will be carried out, including all those patients older than 18 years who go to perform a superior endoscopy with diagnosis of Barrett's esophagus where patients will be randomized into two groups, one of acetic acid and the other of the Seattle protocol as a method Initially and subsequently, a second endoscopy will be performed with the opposite method and the histopathological results of both groups will be compared.
Who Masked: Participant
Masking Description: Participant will be initially allocated in either group without knowing its initial manoeuver
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chromoendoscopy with acetic acid and targeted biopsies (Active Comparator): Acetic acid is prepared at a concentration of 2.5%, after initial cleaning is done, it will be applied with a 7 French spray catheter, starting the proximal application performing a uniform application on the area of intestinal metaplasia an then will be timed for mucous visualization in search of areas of loss of acetowhitening, in case of finding such area will be registered the time in which there was loss of acetowhitening, the distance at which it is located from the upper dental arch in addition to the esophageal face on which the area is located, subsequently evaluation of the glandular pattern is performed only by classifying as normal (glands evenly distributed with normal or abnormal crypt density (compact crypts with increased density; focal irregularity or disorganized crypts; absence of a cryptic pattern), once this evaluation has been carried out, biopsies are directed to these areas to be sent to the pathology service.
  Interventions: Diagnostic Test: Acetic acid chromoendoscopy
- Seattle protocol (Active Comparator): Take random biopsies by quadrants every 2 centimeters biopsy of the intestinal metaplasia areas 1cm above the esophagogastric junction begins, taking tissue every 2cm from the 4 quadrants, separating the biopsies in different bottles based on the length in which they were taken, to later be sent to the pathology service.
  Interventions: Diagnostic Test: Seattle protocol

INTERVENTIONS:
Diagnostic Test: Acetic acid chromoendoscopy — Acetic acid is prepared at a concentration of 2.5% in a 20ml syringe, it will be applied with a 7 french spray catheter compatible with a working channel 2.8mm onwards, starting the proximal application When distally performing a uniform application on the area of intestinal metaplasia and the timed time for mucous visualization in search of areas of loss of acetowhitening begins, in case of finding such area will be registered the time in which there was loss of acetowhitening, the distance at which it is located from the upper dental arch in addition to the face on which the area is located, subsequently evaluation of the glandular pattern is performed only by classifying as normal or abnormal, once this evaluation has been carried out, biopsies are directed to these areas to be sent to the pathology service.
  Arms: Chromoendoscopy with acetic acid and targeted biopsies
Diagnostic Test: Seattle protocol — Take random biopsies by quadrants every 2 centimeters. Biopsy of the intestinal metaplasia areas 1cm above the esophagogastric junction will be initiated, taking tissue every 2cm from the four quadrants, separating the biopsies in different bottles based on the length in which they were taken, to later be sent to the pathology service.
  Arms: Seattle protocol

SUMMARY:
Barrett's esophagus is a complication of chronic gastroesophageal reflux disease that occurs in up to 10% to 15% of patients with this pathology. Well-defined risk factors have been established and are important because they are considered a precancerous lesion (intestinal metaplasia). The conventional diagnostic methods are ineffective in reliably detecting potentially treatable lesions. Investigators propose the use of vital chromoendoscopy with acetic acid using the simplified classification of Portsmouth looking for areas with loss of acetowhitening and taking targeted biopsies to increase the detection of esophageal neoplastic lesions.

DETAILED DESCRIPTION:
Barrett's esophagus is a complication of chronic gastroesophageal reflux disease that occurs in up to 10 to 15% of patients with this disease, well-defined risk factors have been established and are important because they are considered a precancerous condition (metaplasia intestinal). Chromoendoscopy is postulated as an effective way for the detection of esophageal precancerous lesions, early detection and timely treatment with chromoendoscopy with acetic acid being a seemingly reliable alternative, so the investigators will use with the simplified classification of Portsmouth looking for areas with loss of acetowhitening and targeted biopsy to increase the detection of esophageal neoplastic lesions, our main objective being to compare the diagnostic effectiveness of directed biopsies of dysplastic lesions with acetic acid in patients with Barrett's esophagus compared to taking non-directed protocolized biopsies.

A clinical trial will be carried out, including all those patients older than 18 years who go to perform a superior endoscopy with diagnosis of Barrett's esophagus where patients will be up and B Seattle protocol group(four quadrant biopsy every 2 centimeters starting 1 centimeter from above the esophagogastric junction), then proton pump inhibitor washout and crossover allocation with the opposite corresponding manoeuver. Histopathological results of both groups will be compared.

Demographic data of the participants will be collected and the evaluated areas of Barrett's esophagus with each method will be recorded in a data collection sheet detailing in a specific way the number of biopsies taken, specifying if there was loss of acetowhitening and alterations in the mucous pattern and in the case of the opposite arm, the total number of biopsies taken based on the Seattle protocol, said data will be condensed into a database for subsequent statistical analysis and publication of results.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of intestinal metaplasia in follow-up protocol without dysplasia
* Patients whose endoscopic image is suggestive of esophageal intestinal metaplasia and is confirmed by histology
* Barrett's esophagus minimally 2cm
* Patients over 18 years of age who wish to participate in the study
* Signed informed consent

Exclusion Criteria:

* Histological evidence of esophageal adenocarcinoma or known with dysplasia
* History of esophageal ablative therapy
* Known allergy or intolerance to proton pump inhibitors or acetic acid
* Evidence of esophageal varices
* Los Angeles esophagitis C or D
* Uncontrolled coagulopathy (INR> 1.5 or platelets <50,000)
* Pregnancy
* No authorization of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the incidence of dysplasia by directed biopsies with acetic acid chromoendoscopy against taking non-directed protocolized biopsies( Seattle protocol) in patients with Barrett's esophagus. | Patient will be on proton pump inhibitor (PP) for 6-8 weeks
  First the investigators will detect the incidence of dysplasia in Barrett esophagus in patients with acetic acid chromoendoscopy, using the Vienna Classification system by the pathologist.
Comparing the incidence of dysplasia by directed biopsies with acetic acid chromoendoscopy against taking non-directed protocolized biopsies( Seattle protocol) in patients with Barrett's esophagus. | After the wash out time of 6-8 weeks on PPI, this maneuver will be added
  The second maneuver consist on taking non directed biopsies by the Seattle protocol in the same patient. And the incidence of dysplasia on biopsies will be looked for using Vienna Classification system again.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar V Hernandez Mondragon, MD, Principal Investigator — IMSS
Locations (1):
- Centro Medico Nacional Siglo XXI Hospital de Especialidades, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh S, Sharma AN, Murad MH, Buttar NS, El-Serag HB, Katzka DA, Iyer PG. Central adiposity is associated with increased risk of esophageal inflammation, metaplasia, and adenocarcinoma: a systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1399-1412.e7. doi: 10.1016/j.cgh.2013.05.009. Epub 2013 May 22. PMID 23707461
- [Background] Rubenstein JH, Morgenstern H, Appelman H, Scheiman J, Schoenfeld P, McMahon LF Jr, Metko V, Near E, Kellenberg J, Kalish T, Inadomi JM. Prediction of Barrett's esophagus among men. Am J Gastroenterol. 2013 Mar;108(3):353-62. doi: 10.1038/ajg.2012.446. Epub 2013 Jan 15. PMID 23318485
- [Background] Sharma P, Falk GW, Weston AP, Reker D, Johnston M, Sampliner RE. Dysplasia and cancer in a large multicenter cohort of patients with Barrett's esophagus. Clin Gastroenterol Hepatol. 2006 May;4(5):566-72. doi: 10.1016/j.cgh.2006.03.001. Epub 2006 Apr 17. PMID 16630761
- [Background] Shaheen NJ, Falk GW, Iyer PG, Gerson LB; American College of Gastroenterology. ACG Clinical Guideline: Diagnosis and Management of Barrett's Esophagus. Am J Gastroenterol. 2016 Jan;111(1):30-50; quiz 51. doi: 10.1038/ajg.2015.322. Epub 2015 Nov 3. PMID 26526079
- [Background] Chedgy F, Fogg C, Kandiah K, Barr H, Higgins B, McCord M, Dewey A, De Caestecker J, Gadeke L, Stokes C, Poller D, Longcroft-Wheaton G, Bhandari P. Acetic acid-guided biopsies in Barrett's surveillance for neoplasia detection versus non-targeted biopsies (Seattle protocol): A feasibility study for a randomized tandem endoscopy trial. The ABBA study. Endosc Int Open. 2018 Jan;6(1):E43-E50. doi: 10.1055/s-0043-120829. Epub 2018 Jan 12. PMID 29340297
- [Background] Kandiah K, Chedgy FJQ, Subramaniam S, Longcroft-Wheaton G, Bassett P, Repici A, Sharma P, Pech O, Bhandari P. International development and validation of a classification system for the identification of Barrett's neoplasia using acetic acid chromoendoscopy: the Portsmouth acetic acid classification (PREDICT). Gut. 2018 Dec;67(12):2085-2091. doi: 10.1136/gutjnl-2017-314512. Epub 2017 Sep 28. PMID 28970288
- [Background] Tholoor S, Bhattacharyya R, Tsagkournis O, Longcroft-Wheaton G, Bhandari P. Acetic acid chromoendoscopy in Barrett's esophagus surveillance is superior to the standardized random biopsy protocol: results from a large cohort study (with video). Gastrointest Endosc. 2014 Sep;80(3):417-24. doi: 10.1016/j.gie.2014.01.041. Epub 2014 Apr 6. PMID 24713305